CLINICAL TRIAL: NCT05678920
Title: Validation of the Turkish Version of the Modified Early Obstetric Warning Systems (MEOWS) Charts
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Anesthesiologist, Principal Investigator, Samsun Education and Research Hospital
Other Study IDs: MEOWS
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Validation
Keywords: validation; MEOWS; chart; Turkish

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant and postpartum patients: Pregnant patients older than 28th gestational week and patients up to postpartum 6th week who were hospitalized in the obstetrics department
  Interventions: Other: patient-administered questionnaires

INTERVENTIONS:
Other: patient-administered questionnaires — patient-administered questionnaires (MEOWS): Obstetric early warning systems are recommended to provide timely recognition, treatment and early referral of critically ill or developing patients. The development of early warning systems from simple bedside observation charts arose from the knowledge that physiological disturbances precede critical illness. Thanks to these charts, the fact that the patient's findings are in the risky value ranges allows the clinician to evaluate the patient earlier and in detail. MEOWS is a simple screening tool for maternal morbidity.

SUMMARY:
It was aimed to study MEOWS on patients in the obstetrics clinic and to evaluate the performance of this scale as a screening tool and to contribute to its usability in Turkey by translating MEOWS into Turkish.

DETAILED DESCRIPTION:
The Modified Early Obstetric Warning System (MEOWS) is a score-based or color-coded system used to detect changes in physiological parameters and enable earlier recognition and management of deteriorating patients.It was first validated by Sigh et al., then its validity and reliability were demonstrated in many countries, especially in countries with low socio-economic status.Early warning systems are not routinely used in obstetrics clinics in Turkey, and there is no Turkish version of MEOWS in the literature. In this study, it was aimed to study MEOWS on patients in obstetrics clinics and to evaluate the performance of this scale as a screening tool and to validate MEOWS by translating it into Turkish.

The study was carried out in 3 stages. The first stage is the translation of MEOWS into Turkish and its cultural adaptation, the second stage is the use of the study scale and the elimination of deficiencies by conducting a pilot study on 30 patients, and the third stage is the collection and evaluation of patient data until the specified sample size is reached.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients receiving inpatient treatment in obstetrics and gynecology clinics
* Patients whose pregnancy is older than 28 weeks and between 6 weeks postpartum
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients under the age of 18
* Outpatients

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — A study on obstetric patients hospitalized in obstetrics and gynecology clinics.
Study Population: Patients whose pregnancy is older than 28 weeks and between 6 weeks postpartum
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Validation of the Modified Early Obstetric Warning System | Obstetric patients older than 28 weeks of gestation and between 6 weeks postpartum
  Demonstrating the reliability and validity of the Modified Early Obstetric Warning System chart in Turkish. MEOWS chart is contained within a booklet and is commenced on admission to hospital. The same booklet is used during subsequent admissions to hospital during the relevant pregnant and postnatal period. Specific maternal observations that are recorded on the MEOWS chart are diastolic blood pressure, severity of pain, antenatal discharge and/or postnatal lochia and proteinurea. Physiological parameters which deviate from the norm are allocated a score. The score increases as deviation from the norm escalates. The final score then falls into one of three categories: a low, medium, or high score. A low score is 1-4, a medium score is 5-6 and a high score is 7 or more. Any single score of 3 indicates an extreme variation from the normal, which is considered at least a medium score. The colour prompts are green for a low score, amber for medium and red for high scores.
Modified Early Obstetric Warning System Chart | At the end of the study, assessed up to 1 month.
  Calculation of sensitivity, specificity, positive and negative predictive value of the chart

CONTACTS AND LOCATIONS:
Overall Officials: HALE KEFELI CELIK, MD, Study Director — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our data and statistical analysis of each investigated all parameter and data are available after the publication of the clinical study

REFERENCES:
- [Result] Singh S, McGlennan A, England A, Simons R. A validation study of the CEMACH recommended modified early obstetric warning system (MEOWS). Anaesthesia. 2012 Jan;67(1):12-18. doi: 10.1111/j.1365-2044.2011.06896.x. Epub 2011 Nov 9. PMID 22066604
- [Result] Moore J, Thomson D, Pimentil I, Fekad B, Graham W. Introduction of a modified obstetric early warning system -(-MOEWS-)- at an Ethiopian referral hospital: a feasibility assessment. BMJ Open Qual. 2019 Mar 30;8(1):e000503. doi: 10.1136/bmjoq-2018-000503. eCollection 2019. PMID 31206042
- [Result] Tuyishime E, Ingabire H, Mvukiyehe JP, Durieux M, Twagirumugabe T. Implementing the Risk Identification (RI) and Modified Early Obstetric Warning Signs (MEOWS) tool in district hospitals in Rwanda: a cross-sectional study. BMC Pregnancy Childbirth. 2020 Sep 29;20(1):568. doi: 10.1186/s12884-020-03187-1. PMID 32993541
- [Result] Singh A, Guleria K, Vaid NB, Jain S. Evaluation of maternal early obstetric warning system (MEOWS chart) as a predictor of obstetric morbidity: a prospective observational study. Eur J Obstet Gynecol Reprod Biol. 2016 Dec;207:11-17. doi: 10.1016/j.ejogrb.2016.09.014. Epub 2016 Oct 8. PMID 27792988